CLINICAL TRIAL: NCT00199472
Title: Comparison of Dynamic Contrast Enhanced CT and Diuretic Renogram in The Evaluation of Ureteropelvic Junction Obstruction
Brief Title: Comparison of Dynamic Contrast Enhanced CT and Diuretic Renogram in The Evaluation of UPJO
Status: Withdrawn | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: St. Joseph's Health Care London (Other); General Electric (Industry)
Responsible Party: Sponsor
Other Study IDs: 07378
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Ureteral Obstruction
MeSH Terms: conditions — Ureteral Obstruction

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Dynamic Contrast Enhanced CT & Diuretic Renogram

SUMMARY:
Renal blood flow is inversely related to obstruction. We propose that this imaging will be as effective as the diuretic renogram in the functional diagnosis of obstruction. Furthermore, dynamic contrast CT scanning may also add anatomic information necessary for the surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Subjects suspected to have UPJO.

Exclusion Criteria:

* Pregnancy;
* Renal failure (Creatinine >150);
* Allergy to contrast material;
* Ureteral stent;
* Nephrostomy tube;
* Renal pelvis calculi.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Denstedt, MD, FRCSC, Principal Investigator — Urology, St. Joseph's Hospital, University of Western Ontario
Locations (1):
- Urology Clinic, St. Joseph's Hospital, St. Joseph's Health Care London, London, Ontario, Canada